CLINICAL TRIAL: NCT06863571
Title: Reduction of Edema With a Specialized Cocktail for Ultra-early Management in Ischemic Stroke
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RESCUE-IS
Record Dates: First submitted 2025-03-03; First posted 2025-03-07 (Actual); Last update posted 2025-04-18 (Actual); Status verified 2025-02

CONDITIONS: Ischemic Stroke
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- PPA Intervention Group (Experimental): Participants in this group will receive a pharmacological cocktail (PPA) for five days in addition to standard medical treatment for acute ischemic stroke. The regimen includes terazosin or urapidil, and propranolol or esmolol, with individualized blood pressure management. The specific protocol is as follows:
  * Terazosin (no less than 1 mg orally or via nasogastric tube, nightly) or Urapidil (100 mg in 30 mL saline, IV infusion at no less than 2 mL/h)
  * Propranolol (10 mg orally or via nasogastric tube, three times daily) or Esmolol (1 g in 40 mL saline, IV infusion at no less than 2 mL/h; use for no more than 48 hours. Beyond 48 hours, switch to Propranolol)
  Interventions: Drug: PPA Intervention
- Standard Treatment Group (No Intervention): Participants in this group will receive standard medical treatment for acute ischemic stroke without the PPA intervention. This includes appropriate supportive care, blood pressure management according to clinical guidelines, and symptomatic treatment as required.

INTERVENTIONS:
Drug: PPA Intervention — Participants in this group will receive a pharmacological cocktail (PPA) for five days in addition to standard medical treatment for acute ischemic stroke. The regimen includes terazosin or urapidil, and propranolol or esmolol, with individualized blood pressure management. The specific protocol is as follows:
  * Terazosin (no less than 1 mg orally or via nasogastric tube, nightly) or Urapidil (100 mg in 30 mL saline, IV infusion at no less than 2 mL/h)
  * Propranolol (10 mg orally or via nasogastric tube, three times daily) or Esmolol (1 g in 40 mL saline, IV infusion at no less than 2 mL/h; use for no more than 48 hours. Beyond 48 hours, switch to Propranolol)
  Arms: PPA Intervention Group

SUMMARY:
Large ischemic stroke is a severe subtype of acute ischemic stroke (AIS), often leading to malignant cerebral edema, elevated intracranial pressure, and poor functional outcomes. Despite early aggressive treatment, malignant cerebral edema remains a major determinant of prognosis, even in cases of successful recanalization. Preclinical studies suggest that a pharmacological cocktail (PPA) may alleviate cerebral edema by modulating extracellular potassium balance, maintaining aquaporin-4 expression, and enhancing lymphatic drainage.

This multicenter, randomized controlled trial (RCT) aims to assess the safety and efficacy of PPA in reducing cerebral edema and improving outcomes in patients with large ischemic stroke. The study will enroll 68 patients with MCA-territory infarction (80-300 mL infarct volume or ASPECTS 1-5), who are not undergoing decompressive craniectomy. Participants will be randomized to receive PPA therapy or standard treatment. The primary outcome is cerebral edema at 5-7 days, with secondary outcomes including 90-day functional outcomes (mRS) and safety assessments.

DETAILED DESCRIPTION:
Large ischemic stroke is a severe subtype of acute ischemic stroke (AIS), often leading to malignant cerebral edema, elevated intracranial pressure (ICP), and poor functional outcomes. Despite early aggressive treatment, malignant cerebral edema remains a major determinant of prognosis, even in cases of successful recanalization. Patients without endovascular therapy (EVT) also face significant risks of cerebral edema and intracranial hypertension, which contribute to high morbidity and mortality. Preclinical studies suggest that a pharmacological cocktail (PPA) may alleviate cerebral edema by modulating extracellular potassium balance, maintaining aquaporin-4 expression, and enhancing lymphatic drainage. In ischemic stroke models, PPA has demonstrated the potential to accelerate potassium homeostasis and mitigate edema formation, while in traumatic brain injury models, PPA has been shown to promote lymphatic clearance and reduce brain swelling.

This multicenter, randomized controlled trial (RCT) aims to evaluate the safety and efficacy of PPA in reducing cerebral edema in patients with large ischemic stroke. A total of 68 patients with MCA-territory infarction (80-300 mL infarct volume or ASPECTS 1-5) who are not undergoing decompressive craniectomy will be enrolled and randomly assigned to receive PPA therapy or standard treatment in a 1:1 ratio. The primary endpoint is cerebral edema at 5-7 days, assessed by follow-up imaging. Secondary endpoints include functional outcomes at 90 days (mRS) and safety assessments, including adverse events such as hypotension and intracranial hypertension.

The study intervention consists of a PPA regimen over five days, including terazosin or urapidil, and propranolol or esmolol, with individualized blood pressure management based on recanalization status. Imaging and safety monitoring will be conducted throughout the study, and adverse events will be closely tracked and analyzed quarterly. To ensure ethical compliance, informed consent will be obtained from patients or their legally authorized representatives, with mechanisms in place for reconfirmation if the patient regains decision-making capacity. This trial seeks to establish a novel pharmacological approach for cerebral edema management, with the ultimate goal of improving neurological outcomes in large ischemic stroke patients.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Clinical diagnosis of acute ischemic stroke (AIS) in the middle cerebral artery (MCA) territory
* Symptom onset within 3 days (≤72 hours) before randomization
* Infarct volume of 80-300 mL or ASPECTS 1-5 involving at least two cortical regions
* Not scheduled for decompressive craniectomy (either not indicated or declined by the patient/family)
* Written informed consent obtained from the patient or legally authorized representative

Exclusion Criteria:

* Baseline evidence of brain herniation or severe hypotension (SBP <90 mmHg)
* Contraindications to PPA medications (terazosin, urapidil, esmolol, propranolol), such as asthma or severe bradycardia
* Severe comorbidities that may interfere with efficacy assessment or safety monitoring (e.g., end-stage organ failure, advanced malignancy)
* Pregnancy or lactation
* Participation in another interventional trial that may influence study outcomes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Estimated)
Dates: Start 2025-04-12 (Actual); Primary Completion 2026-03-10 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Cerebral Edema at 5-7 Days | 5-7 days post-treatment
  The primary outcome of this study is cerebral edema. Edema will be quantified using standardized imaging analysis techniques. The difference in cerebral edema between the PPA intervention group and the standard treatment group will be compared to evaluate the efficacy of the pharmacological cocktail in reducing brain swelling.

SECONDARY OUTCOMES:
90-Day Functional Outcome (Modified Rankin Scale, mRS) | 90 days post-treatment
  Functional outcomes will be assessed using the modified Rankin Scale (mRS) at 90 days post-treatment, mRS: minimum value = 0, maximum value = 6, and lower scores mean a better outcome
Incidence of Hypotension During the Treatment Period | During the 5-day treatment period
  The occurrence of clinically significant hypotension (defined as systolic blood pressure <90 mmHg) will be monitored throughout the intervention period. The frequency, severity, and need for medical intervention will be compared between the two study groups.
Need for Decompressive Craniectomy | Up to 7 days post-treatment
  The proportion of patients who require decompressive craniectomy (DC) due to worsening cerebral edema and refractory intracranial hypertension will be recorded and compared between the study groups. This will serve as an indicator of treatment efficacy in preventing severe brain swelling.
Mortality at 90 Days | 90 days post-treatment
  All-cause mortality will be recorded and compared between the PPA intervention and standard treatment groups to evaluate the impact of the intervention on survival.
Incidence of Serious Adverse Events (SAEs) | Up to 90 days post-treatment
  All serious adverse events (SAEs), including cardiovascular complications, major bleeding, and severe drug reactions, will be recorded and compared between groups.

CONTACTS AND LOCATIONS:
Locations (1):
- Second Affiliated Hospital of Zhejiang University, School of Medicine, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Undecided